CLINICAL TRIAL: NCT03426852
Title: INVESTIGATING THE EFFECTS SACROILIAC JOINT DYSFUNCTION ON GAIT VARIABILITY IN INDIVIDUALS WİTH LUMBAR HERNIATION NUCLEUS PULPOSUS
Brief Title: INVESTIGATING THE EFFECTS SACROILIAC JOINT DYSFUNCTION ON GAIT IN INDIVIDUALS WITH BACK PAIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, Assoc Prof, Hacettepe University
Other Study IDs: G0-17601
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Biomechanical; Lesion
Keywords: Biomechanical Phenomenon; Gait; Lumbar Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Individuals with lumbar back pain plus sacroiliac disc herniation
  Interventions: Other: No intervention
- Control Group: Individuals with lumbar back pain
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Sacroiliac joint dysfunction (SJD) is a common problem in individuals with lumbar herniation nucleus pulposus (LHNP) plus back pain. It is important to determine the effects of SJD on the gait characteristics in individuals with LHNP.Twelve individuals with LHNP (control group) and six individuals with LHNP plus SJD (study group) will be the participants of the study. Gait characteristics of participants will be evaluate with treadmill. Participants will walk at their self-selected speed for six minutes and data from 2nd minutes to 4th minutes were selected for statistical analyses. Gait speed, cadance, step lengths, time on each foot and step length variabilities will be recorded.

DETAILED DESCRIPTION:
Sacroiliac joint dysfunction (SJD) is a common problem in individuals with lumbar herniation nucleus pulposus (LHNP) plus back pain. It is important to determine the effects of SJD on the gait characteristics in individuals with LHNP.Twelve individuals with LHNP (control group) and six individuals with LHNP plus SJD (study group) will be the participants of the study. Gait characteristics of participants will be evaluate with treadmill. Participants will walk at their self-selected speed for six minutes and data from 2nd minutes to 4th minutes were selected for statistical analyses. Gait speed, cadance, step lengths, time on each foot and step length variabilities will be record

ELIGIBILITY:
Inclusion Criteria:

Have current back pain Have Lumbar Disc Herniation diagnosis Have sacroiliac dysfunction

Exclusion Criteria:

Do not want to participate Have another systemic, neurologic or orthopedic problem

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with lumbar disc herniation with or without sacroiliac dysfunction, age between 18-50 years.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Step Length Variability | First minute
  Covariance of variability for right and left step lenghts.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided